CLINICAL TRIAL: NCT04579380
Title: A Phase 2 Basket Study of Tucatinib in Combination With Trastuzumab in Subjects With Previously Treated, Locally Advanced Unresectable or Metastatic Solid Tumors Driven by HER2 Alterations
Brief Title: Basket Study of Tucatinib and Trastuzumab in Solid Tumors With HER2 Alterations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-019
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Uterine Neoplasms; Uterine Cervical Neoplasms; Biliary Tract Neoplasms; Urologic Neoplasms; Carcinoma, Non-Small-Cell Lung; HER2 Mutations Breast Neoplasms
Keywords: Cervical cancer; Uterine cancer; Biliary tract cancer; Urothelial cancer; Non-squamous non-small cell lung cancer; Non-squamous NSCLC; Breast cancer; Colorectal cancer; Ampullary cancer; Solid tumors; Solid tumors harboring somatic HER2 mutations; Seattle Genetics
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Biliary Tract Neoplasms; Urologic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Colorectal Neoplasms | interventions — tucatinib; Trastuzumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib + Trastuzumab (+ Fulvestrant) (Experimental): Tucatinib + trastuzumab (+ fulvestrant in hormone-receptor positive HER2-mutant breast cancer only)
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: fulvestrant

INTERVENTIONS:
Drug: tucatinib — 300 mg orally twice daily
  Other Names: TUKYSA, ARRY-380, ONT-380
Drug: trastuzumab — Given into the vein (intravenously; IV). 8mg/kg IV on Cycle 1 Day 1, and 6mg/kg every 21 days starting on Cycle 2 Day 1
  Other Names: Herceptin
Drug: fulvestrant — Given into the muscle (intramuscular; IM) once every 4 weeks starting from Cycle 1 Day 1, plus one dose on Cycle 1 Day 15. Only administered to participants with hormone-receptor positive breast cancer.
  Other Names: Faslodex

SUMMARY:
This trial studies how well tucatinib works for solid tumors that make either more HER2 or a different type of HER2 than usual (HER2 alterations) The solid tumors studied in this trial have either spread to other parts of the body (metastatic) or cannot be removed completely with surgery (unresectable).

All participants will get both tucatinib and trastuzumab. People with hormone-receptor positive breast cancer will also get a drug called fulvestrant.

The trial will also look at what side effects happen. A side effect is anything a drug does besides treating cancer.

DETAILED DESCRIPTION:
There are multiple cohorts in this trial:

* 5 tumor specific cohorts with HER2 overexpression/amplification (cervical cancer, uterine cancer, biliary tract cancer, urothelial cancer, and non-squamous non-small cell lung cancer [NSCLC])
* 2 tumor specific cohorts with HER2 mutations (non-squamous NSCLC and breast cancer)
* 2 cohorts which will enroll all other HER2 amplified/overexpressed solid tumor types (except breast cancer, gastric or gastroesophageal junction adenocarcinoma [GEC], and colorectal cancer [CRC]) or HER2-mutated solid tumor types.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of locally-advanced unresectable or metastatic solid tumor, including primary brain tumors
* Participants with non-squamous NSCLC must have progressed during or after standard treatment or for which no standard treatment is available
* Participants with other disease types must have progressed during or after ≥1 prior line of systemic therapy for locally-advanced unresectable or metastatic disease
* Disease progression during or after, or intolerance of, the most recent line of systemic therapy
* Disease demonstrating HER2 alterations (overexpression/amplification or HER2 activating mutations), as determined by local or central testing processed in a Clinical Laboratory Improvement Amendments (CLIA)- or International Organization for Standardization (ISO) accredited laboratory, according to one of the following:

  * HER2 overexpression/amplification from fresh or archival tumor tissue or blood
  * Known activating HER2 mutations detected in fresh or archival tumor tissue or blood
* Have measurable disease per RECIST v1.1 criteria according to investigator assessment
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria

* Participants with breast cancer, gastric or gastroesophageal junction adenocarcinoma, or CRC whose disease shows HER2 amplification/overexpression.
* Previous treatment with HER2-directed therapy; participants with uterine serous carcinoma or HER2-mutated gastric or gastroesophageal junction adenocarcinoma without HER2-overexpression/amplification may have received prior trastuzumab
* Known hypersensitivity to any component of the drug formulation of tucatinib or trastuzumab (drug substance, excipients, murine proteins), or any component of the drug formulation of fulvestrant in participants with HR+ HER2-mutated breast cancer
* History of exposure to a 360 mg/m² doxorubicin-equivalent or >720 mg/m^2 epirubicin-equivalent cumulative dose of anthracyclines
* Treatment with any systemic anti-cancer therapy, radiation therapy, major surgery, or experimental agent within ≤3 weeks of first dose of study treatment or are currently participating in another interventional clinical trial.

There are additional inclusion and exclusion criteria. The study center will determine if criteria for participation are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (103):
- United States (72):
  - HonorHealth, Phoenix, Arizona
  - HonorHealth, Tempe, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope at Huntington Beach, Huntington Beach, California
  - City of Hope at Irvine Sand Canyon, Irvine, California
  - Koman Family Outpatient Pavilion, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UC San Diego Moores Cancer Center- Investigational Drug Services, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope at Long Beach Worsham, Long Beach, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope at Newport Beach Lido, Newport Beach, California
  - City of Hope Torrance, Torrance, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Minnesota Oncology Hematology, PA, Coon Rapids, Minnesota
  - Metro Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - Washington University School of Medicine - Obstetrics & Gynecology [Academic Offices), St Louis, Missouri
  - Barnes-Jewish Hospital Investigational Drug Pharmacy (IDS), St Louis, Missouri
  - Washington University School of Medicine - Obstetrics & Gynecology, St Louis, Missouri
  - Washington University School of Medicine [Patient Clinics], St Louis, Missouri
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - NYU Langone Health - Long Island (Winthrop Hospital), Mineola, New York
  - Perlmutter Cancer Center at NYU Langone GYN Oncology Associates, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center/Duke Cancer Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OSU Wexner Medical Center, CarePoint East, Columbus, Ohio
  - OSU Wexner Medical Center, Ohio State University Hospital East, Columbus, Ohio
  - OSU Wexner Medical Center, Arther G. James Cancer Hospital, and Solove Research Institute, Columbus, Ohio
  - OSU Wexner Medical Center, Investigational Drug Services(IP Ship to), Columbus, Ohio
  - Osu Wexner Medical Center, The Ohio State University Hospital, Columbus, Ohio
  - OSU Wexner Medical Center, Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - OSU Wexner Medical Center, Martha Morehouse Medical Plaza, Columbus, Ohio
  - OSU Wexner Medical Center, OutPatient Care Upper Arlington, Columbus, Ohio
  - OSU Wexner Medical Center, CarePoint Gahanna, Gahanna, Ohio
  - OSU Wexner Medical Center, Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - OSU Wexner Medical Center, Outpatient Care Lewis Center, Lewis Center, Ohio
  - UH Minoff Health Center at Chagrin Highlands, Orange, Ohio
  - OSU Wexner Medical Center, Outpatient Care New Albany, Westerville, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - UPMC Hillman Cancer Center - Washington, Washington, Pennsylvania
  - Prisma Health Cancer Institute, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute, Easley, South Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Prisma Health Cancer Institute, Greer, South Carolina
  - Prisma Health Cancer Institute, Seneca, South Carolina
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hendersonville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Texas oncology-West Texas, Abilene, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - Texas Oncology - Central South, Waco, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - 1 S Park St Medical Center, Madison, Wisconsin
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Belgium (6):
  - Grand Hopital de Charleroi, Charleroi, Hainaut
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Groeninge, Kortrijk
  - CHU de Liege, Liège
  - AZ Sint-Maarten, Mechelen
- Charite Universitatsmedizin Berlin, Berlin, Germany
- Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative lstituto Europeo di Oncologia, Milan, Milan, Italy
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - National Cancer Center Hospital, Cho-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul, Other
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Institut Catala d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Other
  - Cetir Centre Medic, Barcelona
  - Hospital Clínico Universitario de Valencia. Fundación Investigación Clínico de Valencia., Valencia
  - Ascires Eresa Campanar, Valencia
  - Hospital Vithas Valencia 9 de Octubre, Valencia
- United Kingdom (8):
  - Sarah Cannon Research Institute UK, London, Budapest
  - Diagnostic Centre, London, Others
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Guy's Hospital, London
  - Jonathan Poon, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Harley Street Clinic, London
  - Radiology, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okines AFC, Curigliano G, Mizuno N, Oh DY, Rorive A, Soliman H, Takahashi S, Bekaii-Saab T, Burkard ME, Chung KY, Debruyne PR, Fox JR, Gambardella V, Gil-Martin M, Hamilton EP, Monk BJ, Nakamura Y, Nguyen D, O'Malley DM, Olawaiye AB, Pothuri B, Reck M, Sudo K, Sunakawa Y, Van Marcke C, Yu EY, Ramos J, Tan S, Bieda M, Stinchcombe TE, Pohlmann PR. Tucatinib and trastuzumab in HER2-mutated metastatic breast cancer: a phase 2 basket trial. Nat Med. 2025 Mar;31(3):909-916. doi: 10.1038/s41591-024-03462-0. Epub 2025 Jan 17. PMID 39825152
- [Derived] Nakamura Y, Mizuno N, Sunakawa Y, Canon JL, Galsky MD, Hamilton E, Hayashi H, Jerusalem G, Kim ST, Lee KW, Kankeu Fonkoua LA, Monk BJ, Nguyen D, Oh DY, Okines A, O'Malley DM, Pohlmann P, Reck M, Shin SJ, Sudo K, Takahashi S, Van Marcke C, Yu EY, Groisberg R, Ramos J, Tan S, Stinchcombe TE, Bekaii-Saab T. Tucatinib and Trastuzumab for Previously Treated Human Epidermal Growth Factor Receptor 2-Positive Metastatic Biliary Tract Cancer (SGNTUC-019): A Phase II Basket Study. J Clin Oncol. 2023 Dec 20;41(36):5569-5578. doi: 10.1200/JCO.23.00606. Epub 2023 Sep 26. PMID 37751561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with locally-advanced (LA) unresectable or metastatic solid tumors driven by human epidermal growth factor receptor 2 (HER2) alterations, who were previously treated, were enrolled to receive tucatinib in combination with trastuzumab in this study. Participants with hormone-receptor positive breast cancer also received fulvestrant.
Pre-assignment Details: A total of 217 participants were enrolled into 9 separate cohorts based on tumor histology and HER2 alteration status. All 217 participants were treated. Results reported are based on the primary completion date (PCD) of the study; data for only those secondary outcome measures are reported for which analyses were complete at PCD. Remaining outcome measures would be reported upon completion of their analyses at study completion.
Groups:
- Tucatinib+Trastuzumab (Cohort 1): Participants with cervical cancer with HER2 amplification/over expression, received tucatinib 300 milligrams (mg) orally (PO) twice daily (BID) from Day 1 of Cycle 1 onwards and trastuzumab 8 milligram per kilograms (mg/kg) intravenously (IV) on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 2): Participants with uterine cancer with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 3): Participants with biliary tract cancer with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 4): Participants with urothelial cancer with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 5): Participants with non-squamous non-small cell lung cancer (NSCLC) with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 6): Participants with solid tumor types (except breast, gastric or gastroesophageal junction adenocarcinoma [GEC], and colorectal cancer [CRC]) with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 7): Participants with non-squamous NSCLC with HER2 mutations, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8): Participants with breast cancer with HER2 mutations, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants with hormone-receptor positive breast cancer also received fulvestrant 500 mg intramuscular (IM) once every 4 weeks starting from Day 1 of Cycle 1, and on Day 15 of Cycle 1. Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 9): Participants with all solid tumor cancers (except breast and non-squamous NSCLC) with HER2 mutations, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
Period: Overall Study
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9)
Started | 11 | 31 | 30 | 25 | 12 | 31 | 13 | 31 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 31 | 30 | 25 | 12 | 31 | 13 | 31 | 33
Not completed — Death | 9 | 22 | 22 | 17 | 6 | 21 | 10 | 11 | 25
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 0 | 1 | 2 | 0 | 1 | 2
Not completed — Ongoing | 2 | 6 | 4 | 8 | 5 | 8 | 3 | 19 | 6

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were enrolled in the study and received any amount of study treatment.
Groups:
- Tucatinib+Trastuzumab (Cohort 1): Participants with cervical cancer with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 5): Participants with NSCLC with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab (Cohort 6): Participants with solid tumor types (except breast, gastric or GEC, and CRC) with HER2 amplification/over expression, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8): Participants with breast cancer with HER2 mutations, received tucatinib 300 mg PO BID from Day 1 of Cycle 1 onwards and trastuzumab 8 mg/kg IV on Day 1 of Cycle 1 and then 6 mg/kg every 21 days starting on Day 1 of Cycle 2 (1 Cycle = 21 Days). Participants with hormone-receptor positive breast cancer also received fulvestrant 500 mg IM once every 4 weeks starting from Day 1 of Cycle 1, and on Day 15 of Cycle 1. Participants received treatment until unacceptable toxicity, occurrence of radiographic progression or clinical progression, withdrawal of consent, death, or study closure.
- Total: Total of all reporting groups
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9) | Total
Number analyzed (Participants) | 11 | 31 | 30 | 25 | 12 | 31 | 13 | 31 | 33 | 217
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (15.3) | 67.6 (7.4) | 66.4 (10.1) | 67.5 (11.6) | 69.7 (11.1) | 62.7 (10.7) | 71.3 (9.5) | 61.3 (10.3) | 63.8 (10.5) | 64.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 31 | 15 | 6 | 4 | 20 | 6 | 31 | 16 | 140
  Male | 0 | 0 | 15 | 19 | 8 | 11 | 7 | 0 | 17 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 1 | 10
  Not Hispanic or Latino | 11 | 29 | 26 | 17 | 8 | 25 | 9 | 24 | 30 | 179
  Unknown or Not Reported | 0 | 1 | 3 | 6 | 3 | 4 | 4 | 5 | 2 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 9 | 23 | 5 | 3 | 20 | 1 | 11 | 23 | 101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 10
  White | 4 | 18 | 3 | 12 | 6 | 5 | 7 | 15 | 8 | 78
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 6 | 3 | 6 | 4 | 4 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (cORR) as Assessed by Investigator
Description: Confirmed ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version (v)1.1 as assessed by investigator and was considered as confirmed when subsequent response was at least 4 weeks after initial response. As per RECIST v1.1, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeter (mm). PR: at least a greater than or equal to (>=)30 % decrease in the sum of diameters (SOD) of target lesions (longest for non-nodal target lesions and the short axes for nodal target lesions), taking as reference the baseline sum diameters. Disease progression (PD): at least >=20% relative increase in SOD of target lesion taking as reference the smallest sum on study (including baseline sum if that is the smallest on study).
Time Frame: From the first dose of study treatment until the first documented CR or PR on or before the first documented PD or new anti-cancer therapies or death, whichever occurred first (up to 28.3 months)
Population: The Response-Evaluable analysis set includes all participants with measurable disease who meet the following 3 criteria: (1) had a baseline disease assessment, (2) received study treatment, and (3) had post-baseline disease assessment or discontinued treatment due to documented disease progression or clinical progression.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9)
Number analyzed (Participants) | 11 | 30 | 30 | 25 | 12 | 31 | 13 | 31 | 29
Percentage of participants | 27.3 [7.9 to 56.4] | 13.3 [4.7 to 28.0] | 46.7 [30.8 to 63.0] | 8.0 [1.4 to 23.1] | 8.3 [0.4 to 33.9] | 22.6 [11.1 to 38.3] | 0 [0.0 to 20.6] | 41.9 [26.9 to 58.2] | 10.3 [2.9 to 24.6]

2. Secondary Outcome: Confirmed Disease Control Rate (DCR) as Assessed by Investigator
Description: DCR was defined as the percentage of participants with confirmed CR, PR, or stable disease (SD or non-CR/non-PD) according to RECIST v1.1 as assessed by investigator. As per RECIST v1.1, CR: disappearance of all target (T) lesions and non-target (NT) lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least >=30 % decrease in the SOD of target lesions (longest for non-nodal target lesions and the short axes for nodal target lesions), taking as reference the baseline sum diameters. PD: at least >=20% relative increase in SOD of target lesions taking as reference the smallest sum on study (including baseline sum if that is the smallest on study). SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD while on study and cannot have met criteria for PD previously.
Time Frame: From the first dose study treatment until PD or death, whichever occurred first (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

3. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: DOR: time from first documentation of confirmed CR/PR to first documentation of PD according to RECIST v1.1 or death from any cause, whichever occurred earlier. Per RECIST v1.1, CR: disappearance of all T/NT lesions(L). Any pathological lymph nodes (whether T/NT) must have reduction in short axis to <10 mm. PR: at least >=30 % decrease in SOD of TL, taking reference baseline sum diameters. PD: at least >=20% relative increase in SOD of TL taking reference smallest sum on study. Participants who do not have PD & were still on study at time of an analysis/ who have started new anticancer treatment/discontinue prior to documentation of PD were censored at date of last adequate response assessment documenting absence of PD. Participants who had PD/death occurred after two/more consecutive missing scheduled response assessments were censored at date of last adequate response assessment of CR, PR, SD,/non-CR/non-PD. Kaplan-Meier method was used for evaluation.
Time Frame: From the first documented CR or PR until the first documentation of PD or death or censoring date, whichever occurred first (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

4. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by Investigator
Description: PFS was defined as time from the date of treatment initiation to date of PD as per RECIST v1.1 or death from any cause, whichever occurred first . As per RECIST v1.1, PD: least >=20% relative increase in SOD of target lesions taking as reference the smallest sum on study (including baseline sum if that is smallest on study). Participants who do not have PD and were still on study at time of an analysis/ who have started new anticancer treatment/discontinue prior to documentation of PD were censored at date of last adequate response assessment documenting absence of PD. Participants who had PD or death occurred after two or more consecutive missing scheduled response assessments were censored at date of last adequate response assessment of CR, PR, SD,/non-CR/non-PD. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2025-11

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from treatment initiation to death due to any cause. For a participant who was not known to have died by the end of study follow-up, observation of OS was censored on the date the participant was last known to be alive (i.e., the date of last contact). Participants lacking data beyond the day of treatment initiation were censored on the date of treatment initiation (i.e., OS duration of 1 day). Kaplan-Meier method was used for evaluation.
Time Frame: From date of start of study treatment until date of death or censoring date (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. A TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

7. Secondary Outcome: Number of Participants With Treatment Emergent Laboratory Test Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as abnormalities that are new or worsened on or after receiving the first dose of study treatment up to 30 days after the last dose of study treatment. The following laboratory abnormalities were assessed: A-) Hematology: hemoglobin decreased, leukocytes decreased, lymphocytes decreased and increased, neutrophils decreased and platelets decreased; B-) Chemistry: alanine aminotransferase increased, albumin decreased, alkaline phosphatase increased, aspartate aminotransferase increased, calcium corrected for albumin decreased and increased, creatinine increased, glomerular filtration rate estimated decreased, glucose decreased, lactate dehydrogenase increased, magnesium increased and decreased, potassium increased and decreased, sodium increased and decreased and total bilirubin increased.
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: Number of Participants With Any Dose Modifications Due to AEs
Description: Dose modification included dose hold, dose reduction, or discontinuation of drugs. Dose reductions or treatment interruption/discontinuation were made at the discretion of the investigator.
Time Frame: From first dose of the study treatment (Day 1) up to the last dose of study treatment (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Number of Participants With TEAEs of Special Interest
Description: An adverse event of special interest (AESI) were any serious or nonserious AE that were of scientific or medical concern as defined by the sponsor and specific to the program, for which ongoing monitoring and rapid communication to the sponsor were appropriate. A TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab or fulvestrant). AESIs for this study were related to hepatoxicity.
Time Frame: From first dose of the study treatment (Day 1) up to the last dose of study treatment (approximately 52.7 months)
Reporting Status: Not Posted, anticipated posting 2025-11

10. Secondary Outcome: Maximum Concentration (Cmax) of Tucatinib
Time Frame: Cycle 3 Day 1: anytime within 1-4 hours post-dose
Population: The Pharmacokinetic (PK) analysis set included all participants in the safety set from whom at least one evaluable PK assessment was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9)
Number analyzed (Participants) | 11 | 27 | 29 | 22 | 12 | 27 | 13 | 30 | 29
Nanogram per milliliter | 488.2 (104.9) | 483.1 (53.5) | 319.2 (116.2) | 275.9 (122.8) | 437.2 (60.0) | 330.4 (164.2) | 207.7 (344.6) | 393.2 (255.6) | 242.9 (155.1)

11. Secondary Outcome: Trough Concentration (Ctrough) of Tucatinib
Time Frame: Cycle 3 Day 1: Predose
Population: The PK analysis set included all participants in the safety set from whom at least one evaluable PK assessment was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9)
Number analyzed (Participants) | 11 | 27 | 29 | 22 | 12 | 27 | 13 | 30 | 29
Nanogram per milliliter | 196.6 (100.1) | 99.9 (482.9) | 145.7 (383.0) | 105.1 (355.1) | 46.5 (3312.4) | 115.4 (328.3) | 267.4 (165.2) | 126.9 (234.5) | 142.3 (184.1)

ADVERSE EVENTS:
Time Frame: From first dose of the study treatment (Day 1) maximum up to 30 days after the last dose of study treatment death date, or data cut-off date, whichever was earlier (maximum up to 28.8 months)
Description: Same event may appear as both non-serious adverse event and serious adverse event (SAE); however, are presented as distinct events. Event may be categorized as serious in 1 participant and non-serious in another or may have experienced both SAE and non-SAE. Safety analysis set: all participants who received any amount of study drug. All-cause mortality: No. of deaths were reported from Day 1 of study through End of Study for all participants.
Arm/Group | Tucatinib+Trastuzumab (Cohort 1) | Tucatinib+Trastuzumab (Cohort 2) | Tucatinib+Trastuzumab (Cohort 3) | Tucatinib+Trastuzumab (Cohort 4) | Tucatinib+Trastuzumab (Cohort 5) | Tucatinib+Trastuzumab (Cohort 6) | Tucatinib+Trastuzumab (Cohort 7) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) | Tucatinib+Trastuzumab (Cohort 9)
All-Cause Mortality (participants affected / at risk) | 9/11 | 22/31 | 22/30 | 17/25 | 6/12 | 21/31 | 10/13 | 11/31 | 25/33
Serious Adverse Events (participants affected / at risk) | 5/11 | 11/31 | 13/30 | 9/25 | 2/12 | 9/31 | 7/13 | 8/31 | 14/33
Other Adverse Events (participants affected / at risk) | 10/11 | 30/31 | 29/30 | 23/25 | 12/12 | 29/31 | 13/13 | 31/31 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib+Trastuzumab (Cohort 1) (N=11) | Tucatinib+Trastuzumab (Cohort 2) (N=31) | Tucatinib+Trastuzumab (Cohort 3) (N=30) | Tucatinib+Trastuzumab (Cohort 4) (N=25) | Tucatinib+Trastuzumab (Cohort 5) (N=12) | Tucatinib+Trastuzumab (Cohort 6) (N=31) | Tucatinib+Trastuzumab (Cohort 7) (N=13) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) (N=31) | Tucatinib+Trastuzumab (Cohort 9) (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tucatinib+Trastuzumab (Cohort 1) (N=11) | Tucatinib+Trastuzumab (Cohort 2) (N=31) | Tucatinib+Trastuzumab (Cohort 3) (N=30) | Tucatinib+Trastuzumab (Cohort 4) (N=25) | Tucatinib+Trastuzumab (Cohort 5) (N=12) | Tucatinib+Trastuzumab (Cohort 6) (N=31) | Tucatinib+Trastuzumab (Cohort 7) (N=13) | Tucatinib+Trastuzumab+ Fulvestrant (Cohort 8) (N=31) | Tucatinib+Trastuzumab (Cohort 9) (N=33)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (8) | 4 (4) | 7 (13) | 0 (0) | 5 (5) | 2 (2) | 3 (3) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5) | 5 (5) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 4 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 7 (12) | 16 (20) | 12 (18) | 13 (15) | 9 (11) | 13 (19) | 9 (12) | 19 (56) | 12 (14)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (10) | 13 (16) | 6 (6) | 6 (7) | 3 (4) | 7 (7) | 4 (4) | 11 (12) | 9 (10)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (10) | 12 (14) | 4 (6) | 2 (3) | 2 (2) | 7 (10) | 4 (6) | 9 (12) | 10 (13)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 4 (5) | 5 (5) | 7 (7) | 7 (7) | 2 (2) | 11 (12) | 4 (5) | 6 (6) | 13 (13)
Fatigue (General disorders) | 2 (3) | 12 (12) | 4 (4) | 4 (4) | 2 (2) | 5 (5) | 5 (5) | 6 (7) | 7 (7)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (3) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 7 (7) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 4 (5) | 13 (21) | 4 (4) | 1 (1) | 13 (13) | 1 (1) | 6 (8) | 10 (11)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (5)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 5 (5) | 1 (2) | 2 (4) | 3 (3) | 1 (3) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 6 (7) | 8 (8) | 8 (8) | 4 (4) | 12 (13) | 3 (3) | 8 (8) | 12 (12)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 4 (5) | 8 (13) | 5 (6) | 3 (3) | 7 (9) | 3 (5) | 4 (4) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 6 (7) | 4 (4) | 3 (5) | 6 (7) | 2 (2) | 4 (5) | 8 (9)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 5 (6) | 7 (8) | 8 (8) | 5 (6) | 2 (3) | 9 (10) | 3 (4) | 3 (4) | 7 (9)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 3 (3) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 10 (10) | 6 (7) | 4 (4) | 2 (2) | 5 (5) | 3 (3) | 5 (9) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 5 (8) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 4 (5) | 3 (4) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 4 (5) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 7 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 9 (10) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT04579380/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04579380/SAP_001.pdf